CLINICAL TRIAL: NCT05618587
Title: Effect of Low-dose Lithium Therapy on Long COVID Symptoms: a Randomized Controlled Trial.
Brief Title: Effect of Lithium Therapy on Long COVID Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Thomas Guttuso, Professor of Neurology, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00006678; UL1TR001412 (NIH)
Record Dates: First submitted 2022-11-14; First posted 2022-11-16 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Long COVID
Keywords: lithium, long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Lithium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lithium (Experimental): Lithium 10mg po qd
  Interventions: Drug: Lithium
- Placebo (Placebo Comparator): Placebo identically matching the lithium pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium — Lithium has multiple mechanisms of action including anti-inflammatory actions, which may be relevant for treating long COVID.
  Arms: Lithium
Drug: Placebo — Inactive pill
  Arms: Placebo

SUMMARY:
This study will assess low-dose lithium's effects on several different symptoms experienced by long COVID patients.

DETAILED DESCRIPTION:
In this double-blind, placebo-controlled study, 50 patients with long COVID will be randomly assigned to either low-dose oral lithium or placebo therapy for three weeks. After the double-blind study phase, all patients will be provided with lithium therapy for two additional weeks. Study visits will occur at baseline and after the three-week double-blind study phase.

ELIGIBILITY:
1. Documented or self-reported positive test for COVID-19 ≥4 weeks prior to enrollment.
2. No fever for ≥4 weeks prior to enrollment.
3. Reports fatigue and/or brain fog (i.e. concentration or memory impairment) for ≥4 weeks prior to enrollment on the PASC-Specific Symptom questionnaire beginning after infection with COVID-19.
4. Fatigue Severity Scale (FSS) score ≥28 or Brain Fog Severity Scale (BFSS) score ≥28 at baseline.
5. Beck Depression Inventory II score <24.
6. No change in any psychoactive or steroid medications for ≥30 days.
7. No plan to change any psychoactive, steroid or diuretic medication for ≥5 weeks and not planning on obtaining a COVID vaccine within the next 5 weeks.
8. Not using any long COVID therapies felt to be worsening the patient's symptoms or starting a long COVID therapy within the next 5 weeks.
9. No history of fibromyalgia, chronic fatigue syndrome or progressive cognitive disorder prior to COVID-19 infection.
10. No active medical, psychiatric or social problems that would interfere with completing the study procedures in the opinion of the investigator.
11. No use of tobacco or marijuana products for >6 months and no current alcohol abuse (≥4 drinks/day) or illicit drug use.
12. Not receiving or applying for disability payments or workman's compensation for long COVID.
13. Not pregnant or nursing or planning to get pregnant over the next two months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Guttuso, Jr., MD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Williamsville, New York, United States

REFERENCES:
- [Derived] Guttuso T Jr, Zhu J, Wilding GE. Lithium Aspartate for Long COVID Fatigue and Cognitive Dysfunction: A Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2436874. doi: 10.1001/jamanetworkopen.2024.36874. PMID 39356507

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lithium | Placebo
Started | 26 | 26
Completed | 24 | 26
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium | Placebo | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 20 | 33
  >=65 years | 11 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (14.3) | 55.0 (13.7) | 58.5 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 22 | 26 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 26 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Severity Scale
Description: 7-item questionnaire assessing fatigue severity. Score range 1-49 with higher values signifying worse outcome
Time Frame: Change from baseline to day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
score on a scale | -11.3 (12.6) | -8.6 (12.3)
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 0.46, t-test, 2 sided

2. Primary Outcome: Brain Fog Severity Scale
Description: 7-item questionnaire assessing brain fog severity. Score range 1-49 with higher values signifying worse outcome
Time Frame: Change from baseline to day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
score on a scale | -9.0 (13.8) | -8.1 (10.6)
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 0.79, t-test, 2 sided

3. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Change in symptoms on 7-point scale. Single-item scale. Score range 1-7 with higher values signifying better outcome
Time Frame: Day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
score on a scale | 4.7 (1.1) | 4.6 (1.2)
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 0.68, t-test, 2 sided

4. Secondary Outcome: Well-Being Scale
Description: Sense of well-being over past week on 10-point scale. Score range 0-10 with higher values signifying better outcome.
Time Frame: Change from baseline to day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
score on a scale | 1.0 (2.0) | 0.9 (2.1)
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 0.89, t-test, 2 sided

5. Secondary Outcome: Short Form-12 Health Survey (1-week Modification)
Description: Quality of life assessment over past week, PCS-subscale. 12-item quality of life scale. Score range 0-100 for both the Physical Component Score and the Mental Component Score with higher values signifying better outcomes.
Time Frame: Change from baseline to day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
score on a scale | 5.1 (8.5) | 4.2 (11.1)
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 0.75, t-test, 2 sided

6. Secondary Outcome: Desire to Continue Therapy
Description: Single Yes/No question. Single-item scale. Score range 1-2 with higher value signifying better outcome. Reported as % of respondents recording "yes".
Time Frame: Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
Participants | 12 | 13
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 1.0, Barnard unconditional exact test

7. Secondary Outcome: Generalized Anxiety Disorder-2 Scale
Description: 2-item questionnaire assessing anxiety frequency over the past week. 2-item scale. Score range 0-6 with higher values signifying worse outcome
Time Frame: Change from baseline to day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
score on a scale | -0.8 (1.7) | -1.4 (1.7)
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 0.28, t-test, 2 sided

8. Secondary Outcome: Headache and Body Pain Bother Scale
Description: 2-item questionnaire assessing frequency of headaches and body pain over the past week, Headache score. 2-item scale. Score range 2-10 with higher values signifying worse outcome
Time Frame: Change from baseline to day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
score on a scale | -0.6 (0.7) | -0.7 (1.2)
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 0.58, t-test, 2 sided

9. Secondary Outcome: Insomnia Severity Index
Description: 7-item questionnaire assessing insomnia severity over the past week. 7-item scale. Score range 0-28 with higher values signifying worse outcome.
Time Frame: Change from baseline to day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
score on a scale | -6.0 (6.7) | -4.4 (4.8)
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 0.41, t-test, 2 sided

10. Secondary Outcome: Sense of Smell and Taste Change Scale
Description: Subjective change from baseline on a 7-point scale (score range: 1-7) with higher scores indicating better outcomes. Scores of 1 and 7 indicate sense of smell and taste were "very much worse" or "very much improved", respectively, since the start of study treatment.
Time Frame: Day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
score on a scale | 4.1 (0.3) | 4.2 (0.4)
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 0.50, t-test, 2 sided

11. Secondary Outcome: Digit Symbol Substitution Test
Description: Validated cognitive test. Score range 0-100 with higher scores indicating a better outcome.
Time Frame: Change from baseline to day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
score on a scale | 4.3 (5.9) | 6.6 (9.0)
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 0.29, t-test, 2 sided

12. Secondary Outcome: Delayed Recall Test
Description: Validated cognitive test. Score range 0-5 with higher scores indicating better outcomes.
Time Frame: Change from baseline to day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium | Placebo
Number analyzed (Participants) | 24 | 26
score on a scale | 0.46 (1.02) | 0.35 (0.80)
Statistical Analysis 1: Comparison: Lithium vs Placebo; Test type: Superiority; p = 0.35, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 5-weeks
Arm/Group | Lithium | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT05618587/Prot_SAP_000.pdf